CLINICAL TRIAL: NCT01536873
Title: A Dolutegravir Open Label Protocol for HIV Infected, Adult and Adolescent Patients With Integrase Resistance
Brief Title: Dolutegravir Expanded Access Study
Acronym: DEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114916; 2011-001646-16 (EudraCT Number)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: treatment experienced patients; Integrase resistance
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dolutegravir — Eligible patients will receive DTG 50 mg given orally BID

SUMMARY:
ING114916 is an open-label, multi-center, expanded access (EAP) study

DETAILED DESCRIPTION:
ING114916 is an open-label, multi-center EAP to allow access to patients with HIV-1 infection who have documented raltegravir or elvitegravir resistance, have limited treatment options and require dolutegravir to construct a viable anti-retroviral regimen for therapy. Patients must not be eligible for another ongoing dolutegravir clinical trial in order to participate in this EAP.

The duration of patient accrual into the study will extend until dolutegravir receives local (by country) regulatory approval.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects greater than 18 years of age 2. Documented HIV-1 RNA >/= 400 c/mL 3. Documented raltegravir or elvitegravir resistance 4. Inability to construct a viable background ART regimen with commercially available medications.

-

Exclusion Criteria:

1. Creatnine clearance < 30ml/min via Cockcroft-Gault method
2. Females who are pregnant and/or breastfeeding
3. Patients with known integrase allergic reaction
4. ALT > 5 times the ULN within one month of treatment initiation
5. ALT > 3 times ULN and total bilirubin >1.5 times ULN
6. Evidence of severe hepatic impairment
7. Patients eligible for, and have access to, an actively enrolling DTG Phase III clinical study
8. Any condition or any active clinically significant disease during screening, anticipated requirement for any prohibited concomitant medications -

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06-14 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Expanded access | Not applicable for an expanded access study
  To to provide access in an open label protocol program to patients who have documented RAL or ELV resistance, who have limited treatment options and who require DTG to construct a viable ARV regimen for therapy

SECONDARY OUTCOMES:
Assess adverse events | Not applicable for an expanded access study
  Assess any serious adverse events (SAEs) and adverse events (AEs) that lead to the discontinuation of DTG 50 mg BID

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (61):
- United States (20):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
- Austria (3):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
- Brazil (10):
  - GSK Investigational Site, Ipanema, Rio de Janeiro
  - GSK Investigational Site, Macaé, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Fortaleza
  - GSK Investigational Site, Maceió
  - GSK Investigational Site, Ribeirão Preto
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vittoria
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- Germany (8):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Mannheim
- Italy (7):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Venezia
- GSK Investigational Site, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided